CLINICAL TRIAL: NCT03366506
Title: Investigation of the Epidemiological Factors Associated With the Development of Amyotrophic Lateral Sclerosis (ALS)
Acronym: EpidALS
Status: Recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0633-08-HMO-CTIL
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: ALS
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALS patients: ALS patients ( suspected, possible, probable or definite per El-Escorial criteria).
  Observation
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
Investigation of the epidemiological factors associated with amyotrophic lateral sclerosis (ALS) in Israel with a view to future international collaboration. Particularly addressing:-

1. Differences between ethnic subgroups
2. Differences between immigrant and native-born populations
3. Differences according to military service profile Clinical features gathered at each routine visit ,throughout the entire course of the disease, will be recorded in database format, in order to correlate with potential epidemiological factors.

DETAILED DESCRIPTION:
Investigation of the epidemiological factors associated with amyotrophic lateral sclerosis (ALS) in Israel with a view to future international collaboration. Particularly addressing:-

1. Differences between ethnic subgroups
2. Differences between immigrant and native-born populations
3. Differences according to military service profile Clinical features gathered at each routine visit ,throughout the entire course of the disease, will be recorded in database format, in order to correlate with potential epidemiological factors.

The clinical features will include pattern of onset, details of full clinical exam ( including ALSFRS-R score, power, reflexes, and other signs of upper or lower-motor neuron dysfunction.

Correlations between different clinical parameters themselves will be made, as well as correlation between clinical parameters and other epidemiological factors.

ELIGIBILITY:
Inclusion Criteria:

- Suspected, possible, probable ,definite ALS

Exclusion Criteria:

-

Ages: 12 Years to 120 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Population referred to ALS clinic with suspected, possible, probable ,definite ALS
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-03-09 (Actual); Primary Completion 2049-03 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
Progression rate | up to 10 years
  Progression of ALSFRS-R score over time

SECONDARY OUTCOMES:
Appearance of clinical features of UMN or LMN dysfunction | 10 years
  Appearance of clinical features of UMN or LMN dysfunction over time

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gotkine, MBBS, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organisation, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Via specific collaboration agreements.